CLINICAL TRIAL: NCT05794139
Title: A Phase 2, Randomised, Double-blind, Placebo-controlled, 2-way Crossover Study to Evaluate the Efficacy, Safety, and Tolerability of NMD670 in Ambulatory Adults With Type 3 Spinal Muscular Atrophy
Brief Title: Safety and Efficacy of NMD670 in Ambulatory Adult Patients With Type 3 Spinal Muscular Atrophy
Acronym: SYNAPSE-SMA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: NMD Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NMD670-02-0001; 2022-002301-24 (EudraCT Number)
Record Dates: First submitted 2023-03-15; First posted 2023-04-03 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Spinal Muscular Atrophy
Keywords: Transmission Enhancer; Neuromuscular Junction Transmission; ClC-1
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Intervention Model Description: 2-way crossover
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental): Experimental drug followed by placebo
  Interventions: Drug: NMD670; Drug: Placebo
- Cohort 2 (Experimental): Placebo followed by experimental drug
  Interventions: Drug: NMD670; Drug: Placebo

INTERVENTIONS:
Drug: NMD670 — Tablets
Drug: Placebo — Tablets

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, tolerability and pharmacokinetics of NMD670 in the treatment of ambulatory adults with spinal muscular atrophy type 3

ELIGIBILITY:
Inclusion Criteria:

1. Participants with a clinical diagnosis of Type 3 SMA.
2. Participants who are ambulatory, defined as being able to walk at least 50 metres without walking aids at screening during the 6-minute walk test.
3. Participant with genetic confirmation of diagnosis (e.g., homozygous deletion or compound heterozygous deletion and mutation of survival of motor neuron 1 gene [SMN1])
4. Participant with 3 to 5 copies of survival of motor neuron 2 gene [SMN2].
5. Participant has a body mass index (BMI) within the range 19-35 kg/m2 (inclusive).
6. Participant is male or female.
7. Contraceptive use by men and women must be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
8. Participant is capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in the protocol.

Exclusion Criteria:

1. Participants with prior surgery or fixed deformity (scoliosis, contractures) which would restrict ability to perform study-related tasks.
2. Participants with other significant disease that may interfere with the interpretation of study data (e.g., other neuromuscular or muscular diseases).
3. Participants with other significant clinical and/or laboratory safety findings that may interfere with the conduction or interpretation of the study
4. Participants received treatment with an investigational medical product (IMP) within 30 days (or 5 half-lives of the medication, whichever is longer) prior to Day 1.
5. Participants with history of poor compliance with relevant SMA therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-09-21 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in 6 minute walk test (6MWT) total distance versus placebo | Baseline to day 21
  Distance walked (meters)

SECONDARY OUTCOMES:
Change from baseline in muscle strength versus placebo | Baseline to day 21
  Handgrip, knee flexor, elbow flexor, elbow extension and should abduction (Newton)
Change from baseline in 6 minute walk test (6MWT) fatigue index versus placebo | Baseline to day 21
  percentage change in distance walked in 6th minute compared to 1st minute
Change from baseline in Revised Hammersmith Scale (RHS) versus placebo | Baseline to day 21
  Total score. Scale goes from 0-69 and higher score indicates improvement of symptoms
Change from baseline in jitter versus placebo | Baseline to day 21
  Jitter (micro seconds) assessed with single fiber EMG
Change from baseline in blocking versus placebo | Baseline to day 21
  Blocking (%) assessed with single fiber EMG
Incidence of treatment emergent adverse events | Over 21 days of dosing
  Summarised per treatment
Incidence of serious treatment emergent adverse events | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on physical examinations | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on safety laboratory parameters | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant vital signs abnormalities | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant ECG abnormalities | Over 21 days of dosing
  Summarised per treatment
Incidence of Suicidal Ideation or Suicidal Behavior | Over 21 days of dosing
  Summarised per treatment
Incidence of clinically significant abnormalities on opthalmological examinations | Over 21 days of dosing
  Summarised per treatment

CONTACTS AND LOCATIONS:
Locations (29):
- United States (10):
  - UCLA David Geffen School Of Medicine - Neurology, Los Angeles, California
  - Stanford University Medical Center, Palo Alto, California
  - UF Fixel Institute for Neurological Diseases, Gainesville, Florida
  - Rare Disease Center, Atlanta, Georgia
  - University of Kansas Medical Center, Kansas City, Kansas
  - Roy Blunt NextGen Precision Health Institute, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Rare Disease Research - Raleigh-Durham, Hillsborough, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Neurology Rare Disease Center, Denton, Texas
- Belgium (2):
  - UZ Leuven - Neurochirurgie Campus Gasthuisberg, Leuven
  - CHR de la Citadelle - Neurologie, Liège
- Canada (2):
  - Heritage Medical Research Clinic, Calgary
  - Genge Partners Inc., Montreal
- Denmark (2):
  - Aarhus Universitetshospital, Neurologisk Afdeling, Aarhus
  - Rigshospitalet - Neurologisk Afdeling, Copenhagen
- Germany (2):
  - Charite - Campus Virchow-Klinikum (CVK), Berlin
  - Universitätsklinikum Essen - Klinik Für Neurologie, Essen
- Italy (6):
  - Istituto Giannina Gaslini, IRCCS, Genova
  - Istituto Neurologico C. Besta, Fondazione IRCCS, Milan
  - Ospedale Niguarda, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Università degli studi di Pisa, Pisa
  - PU A. Gemelli, Università Cattolica del Sacro Cuore, Roma
  - AOU Città della Salute e della Scienza di Torino, Torino
- Universitair Medisch Centrum Utrecht, locatie Academisch Zie - Neurology, Utrecht, Netherlands
- Spain (4):
  - Hospital Universitari Vall D Hebron, Barcelona
  - H. Donostia, Donostia / San Sebastian
  - Hospital Materno Infantil La Paz, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No